CLINICAL TRIAL: NCT06483893
Title: Comparison of Ultrasound-Guided Thyroid Cartilage Plane Block and Ultrasound-Guided Traditional Superior Laryngeal Nerve Block for Awake Fiberoptic Intubation in Patients With Limited Neck Mobility Undergoing Cervical Spine Fixation
Brief Title: Ultrasound-Guided Thyroid Cartilage Plane Block vs Ultrasound-Guided Traditional Superior Laryngeal Nerve Block for Awake Fiberoptic Intubation in Patients With Limited Neck Mobility Undergoing Cervical Spine Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/04062024/Fakhry
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Patient Satisfaction
Keywords: Thyroid Cartilage; Awake Fiberoptic Intubation; Cervical Spine; Superior Laryngeal Nerve
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thyroid cartilage plane block group (TCPB Group) (Active Comparator): Participants in the (group TCPB) will receive US-guided thyroid cartilage plane block. Ultrasound-guided bilateral Thyroid Cartilage Plane Block is performed using the thyroid cartilage plate as an anatomical landmark. 3ml of 2% lidocaine is injected on the surface of the thyroid cartilage plate. Subsequently, perform fiberoptic bronchoscope-guided oropharyngeal, subglottic, and tracheal surface anesthesia. After completing surface anesthesia, perform fiberoptic bronchoscope-guided tracheal intubation, securing it properly.
  Interventions: Procedure: US-guided thyroid cartilage plane block (group TCPB)
- traditional superior laryngeal nerve block group (Traditional SLNB Group) (Active Comparator): Participants in the (group traditional SLNB) will receive US-guided traditional superior laryngeal nerve block. Traditional Superior Laryngeal Nerve Block is performed using the thyrohyoid muscle and thyrohyoid membrane as an anatomical landmark. The thyroid cartilage and the greater horn of hyoid bone are hyperechoic signals on sonography. 3ml of 2% lidocaine is injected above the thyrohyoid membrane next to the superior laryngeal artery between two hyperechoic structures. Subsequently, perform fiberoptic bronchoscope-guided oropharyngeal, subglottic, and tracheal surface anesthesia. After completing surface anesthesia, perform fiberoptic bronchoscope-guided tracheal intubation, securing it properly.
  Interventions: Procedure: US-guided traditional superior laryngeal nerve block (group traditional SLNB)

INTERVENTIONS:
Procedure: US-guided thyroid cartilage plane block (group TCPB) — Participants in the (group TCPB) will receive US-guided thyroid cartilage plane block. Ultrasound-guided bilateral Thyroid Cartilage Plane Block is performed using the thyroid cartilage plate as an anatomical landmark. 3ml of 2% lidocaine is injected on the surface of the thyroid cartilage plate. Subsequently, perform fiberoptic bronchoscope-guided oropharyngeal, subglottic, and tracheal surface anesthesia. After completing surface anesthesia, perform fiberoptic bronchoscope-guided tracheal intubation, securing it properly.
  Arms: thyroid cartilage plane block group (TCPB Group)
Procedure: US-guided traditional superior laryngeal nerve block (group traditional SLNB) — Participants in the (group traditional SLNB) will receive US-guided traditional superior laryngeal nerve block. Traditional Superior Laryngeal Nerve Block is performed using the thyrohyoid muscle and thyrohyoid membrane as an anatomical landmark. The thyroid cartilage and the greater horn of hyoid bone are hyperechoic signals on sonography. 3ml of 2% lidocaine is injected above the thyrohyoid membrane next to the superior laryngeal artery between two hyperechoic structures. Subsequently, perform fiberoptic bronchoscope-guided oropharyngeal, subglottic, and tracheal surface anesthesia. After completing surface anesthesia, perform fiberoptic bronchoscope-guided tracheal intubation, securing it properly.
  Arms: traditional superior laryngeal nerve block group (Traditional SLNB Group)

SUMMARY:
The aim of the work to compare between the effectiveness and safety of ultrasound-guided superior laryngeal nerve block through surface injection of local anesthetic solution on the thyroid cartilage and ultrasound-guided traditional superior laryngeal nerve block on quality of airway anesthesia for awake fiberoptic intubation in patients with limited neck mobility undergoing cervical spine fixation.

DETAILED DESCRIPTION:
The difficult airway is a challenge for the anesthesiologist. When a patient presents with anticipated difficult airway, the strategies can be varied, depending on the clinical context, the available resources, and the level of training of human resources. However, most clinical practice guidelines agree that difficult airway management shall be approached with the patient awake. Intubating the patient awake improves the perioperative safety, since it allows for spontaneous breathing, maintaining the patency of the airway, and cooperation with the operator.

Awake fibreoptic intubation (AFOI) is the gold standard in the management of the difficult airway.

Several ways to administer local anaesthetic to the upper airway to aid AFOI have been described including nebulisation, spray-as-you-go techniques and airway nerve blocks, each with its own potential advantages and disadvantages.

The objective of the ideal technique is the use of the lowest possible dose of the local anesthetic agent, to achieve a successful block that facilitates the intubation conditions, and increases the safety and tolerability of the patient.

Airway topicalization is commonly used to facilitate awake tracheal intubation and can be implemented in various ways. There are reservations about performing topical anesthesia of the airway because of some unsolved drawbacks, including poor airway anesthesia quality due to unreliable effects and the increased risk of exceeding the maximum dose of local anesthesia, leading to local anesthetic systemic toxicity (LAST).

Airway nerve blocks provide better anesthesia quality for awake tracheal intubation and lower overall complications than topical anesthesia.

Ultrasound-guided superior laryngeal nerve block is a viable alternative for topical anesthesia during awake tracheal intubation. However, direct recognition of the superior laryngeal nerve under ultrasonography can be challenging due to its small dimensions and large probe size. Several methods have been reported to block the superior laryngeal nerve, utilizing the thyroid hyoid membrane and superior laryngeal artery as anchors to locate the superior laryngeal nerve.

Thyroid cartilage plane block is a new approach for local anesthetic injection targeting an interfascial plane between the thyroid cartilage laminae and the muscle groups above. This approach, distant from any nerves or vascular structures, may offer enhanced safety compared to the superior laryngeal nerve space block.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18-65 years
* either gender
* ASA I-II
* limited neck mobility

Exclusion Criteria:

* patients who refuse to give consent
* non-cooperative patients
* have asthma or ischemic heart disease
* preoperative hoarseness, sore throat
* mental or neurological disorders
* contraindications for regional block (coagulopathy , infection at the needle insertion site and allergy to local anesthetics)
* body mass index (BMI) >26 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
the time taken to perform block | During surgery, upon performing block
  from the start of ultrasound probe positioning to completion of drug administration

SECONDARY OUTCOMES:
quality of airway anesthesia a | During surgery, upon intubation
  Assessment of quality of airway anesthesia was done on a 5-point scale as described by Reasoner et al.[13] 0 = No coughing or gagging in response to intubation, 1 = Mild coughing and/or gagging that did not hinder intubation, 2 = Moderate coughing and/or gagging that interfered minimally with intubation, 3 = Severe coughing and/or gagging that made intubation difficult, 4 = very severe coughing and/or gagging that required additional local anesthetic (LA) and/or change in technique to achieve successful intubation.
Ramsay Sedation Score | T0: upon entry to the operating room,T1: before insertion of the tracheal tube,T2: immediately after tracheal tube insertion,T3: 5 minutes after successful intubation ]
  The Ramsay Sedation Score is as follows: 6 points for unarousable, 5 points for slow response to stimulus, 4 points for asleep but easily aroused, 3 points for quiet and cooperative with orientation, 2 points for asleep, anxious, restless, and 1 point for asleep, agitated, and restless. Satisfactory sedation falls within 2-4 points, while oversedation is indicated by 5-6 points.

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University hospital, Banī Suwayf, Beni Suweif Governorate, Egypt